CLINICAL TRIAL: NCT00794066
Title: Prevalence of Peripheral Arterial Disease in Acute Ischemic and Hemorrhagic Stroke Patients
Brief Title: Peripheral Arteriopathy Rate In Stroke
Acronym: PARIS
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: PARIS-Study2009
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Artery Disease
Keywords: PAD; Stroke; ICH; prevalence
MeSH Terms: conditions — Peripheral Arterial Disease; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: TIA
  Interventions: Procedure: measuring the ankle brachial index
- 2: Ischemic stroke
  Interventions: Procedure: measuring the ankle brachial index
- 3: Hemorrhagic stroke
  Interventions: Procedure: measuring the ankle brachial index

INTERVENTIONS:
Procedure: measuring the ankle brachial index — Assessment of the ankle brachial index using the "boso-ABI-system 100" (www.boso.de).

SUMMARY:
Purpose:

To assess the prevalence of peripheral arterial disease (PAD) in acute stroke patients.

Interventions:

Assessment of the ankle brachial index using the "boso-ABI-system 100" (www.boso.de).

Design:

Prospective, open, cohort study.

Study size planned:

1500.

Follow-up duration:

3 months.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients with acute ischemic or hemorrhagic stroke.

Exclusion Criteria:

* Congestive heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with acute ischemic or hemorhagic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2008-08; Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Functional outcome (modified Rankin Scale) | 3 months

SECONDARY OUTCOMES:
Prevalence of peripheral arterial disease | during hospital stay
  Presence or not of PAD as assessed using ABI during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwab, MD, Study Director — Head of the Department of Neurology, University of Erlangen, Germany
Locations (1):
- Department of Neurology, University of Erlangen, Germany, Erlangen, Germany